CLINICAL TRIAL: NCT03290560
Title: A Randomized, Double-blind, Placebo-controlled Phase II Multi-Center Evaluation to Assess the Safety and Tolerability of DM199 Administered Intravenously and Subcutaneously in Subjects With Acute Ischemic Stroke
Brief Title: Evaluation to Assess Safety and Tolerability of DM199 in Subjects With Acute Ischemic Stroke
Acronym: ReMEDy1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DiaMedica Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DM199-2017-001
Record Dates: First submitted 2017-09-18; First posted 2017-09-25 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2020-02

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — DM199

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Recombinant human tissue kallikrein (Experimental): A single IV infusion of 1 microgram/kg followed by 8 subcutaneous injections of 3 microgram/kg occurring every 72 hours.
  Interventions: Drug: Recombinant human tissue kallikrein
- Placebo (Placebo Comparator): A single IV infusion of 1 microgram/kg followed by 8 subcutaneous injections of 3 microgram/kg occurring every 72 hours.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Recombinant human tissue kallikrein — Recombinant human tissue kallikrein
  Other Names: DM199
  Arms: Recombinant human tissue kallikrein
Other: Placebo — Placebo Comparator: Phosphate buffered saline
  Arms: Placebo

SUMMARY:
This is a Phase II study to assess the safety and tolerability of DM199 in acute ischemic stroke patients. The study will be randomized, placebo controlled at multiple centers.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is >/= 18 years of age
2. Subject has been diagnosed with acute ischemic stroke with onset ≤ 24 hours from enrollment.
3. Subject has NIH stroke score (NIHSS) ≥ 6 and ≤ 25.
4. Subject or legally authorized representative is willing and able to sign written informed consent.

Exclusion Criteria:

1. Subject is currently prescribed angiotensin-converting-enzyme inhibitors (ACEi) and is unable or unwilling to convert to another antihypertensive pharmacological treatment during the active treatment period (+5 days) of the study.
2. Subject has a history of significant allergic diathesis such as urticaria, angioedema or anaphylaxis.
3. Subjects with current malignancy or active malignancy ≤ 3 years prior to enrollment except basal cell or squamous cell carcinoma of the skin or in situ cervical cancer that has undergone potentially curative therapy and at least six months have elapsed since the procedure.
4. Subject has a history of clinically significant acute bacterial, viral, or fungal systemic infections in the last four weeks prior to enrollment.
5. Subject has clinical or laboratory evidence of an active infection at the time of enrollment.
6. Subject has known alpha 1-antitrypsin deficiency (α1-antitrypsin deficiency).
7. Subject has a known diagnosis of human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or anti-hepatitis C virus (Anti-HCV) at screening.
8. Subject is pregnant or nursing.
9. Subject is male or female of childbearing potential, is participating in heterosexual sexual activity that could lead to pregnancy, and is unable or unwilling to practice medically effective contraception during the study.
10. Subject is participating in any other investigational device or other drug study ≤ 4 weeks or 5 half-lives of the investigational product, whichever is longer.
11. Subject does not have sufficient venous access for infusion of study treatment or blood sampling.
12. In the opinion of the Investigator, subject is unlikely to be followed for the duration of t the study.
13. Subject is unable or unwilling to comply with protocol requirements, including assessments, tests, and follow-up visits.
14. Subject has any other medical condition which in the opinion of the Investigator will make participation medically unsafe or interfere with the study results.
15. Pre-stroke Modified Rankin Scale ≥4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.3 | 90 Days
  Assessed by total number and severity of all treatment-related adverse events.

SECONDARY OUTCOMES:
Changes from baseline to Day 90 of NIH Stroke Scale. | 90 Days
  Assessed by a reduction in points from baseline.
Changes from baseline to Day 90 of Barthel Index. | 90 Days
  Assessed by an increase in points from baseline.
Changes from baseline to Day 90 of Modified Rankin Scale. | 90 Days
  Assessed by a reduction in points from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Campbell, Principal Investigator — Melbourne Health
Locations (12):
- Australia (12):
  - Lismore Base Hospital, Lismore, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Princess Alexandria Hospital, Woolloongabba, Queensland
  - Alfred Health, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Sunshine Hospital, St Albans, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Royal Adelaide Hospital, Adelaide
  - Ballarat Health Services, Ballarat
  - Box Hill Hospital, Box Hill

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Campbell BC, Kasner SE, Lista AD, Volpi JJ, Kleinig TJ, Cordato D, Dewey HM, Choi PM, Garcia-Esperon C, Sahathevan R, Wijeratne T, Wong AA, Ghia D, Cloud GC, Giuffre M, Bath PM; ReMEDy1 Investigators. Safety and tolerability of Rinvecalinase Alfa (DM199) for acute ischemic stroke (ReMEDy1). Int J Stroke. 2025 Nov 6:17474930251396480. doi: 10.1177/17474930251396480. Online ahead of print. PMID 41195862

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT03290560/Prot_SAP_000.pdf